CLINICAL TRIAL: NCT07079774
Title: Post-Market Clinical Follow-up Study of the TrueLok Elevate Transverse Bone Transport System for the Treatment of Lower Limb Ulcers as Soft Tissue Defects
Brief Title: TrueLok Elevate PMCF Study
Status: Recruiting | Type: Observational
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-TLEL-25
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Wound of Skin; Ulcers; Soft Tissue Defect
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transverse Bone Transport System — This is a prospective, international, multicentre, observational post-market clinical follow-up (PMCF) study. Adult subjects will be treated according to the manufacturer's Instructions for Use, with follow-up extending to 12 months post-device removal. Participating sites include centres in the US, Europe, the UK, and South Africa.
  Subjects will be followed using a phased framework:
  T0: Index Surgery (baseline data, operative details, ulcer status) T1: End of Distraction (device parameters, adverse events, ulcer status) T2: End of Compression (similar to T1) T3: Device Removal (confirmation of union, ulcer status)
  Post-removal visits:
  F3: 3 months F6: 6 months F12: 12 months

SUMMARY:
The TrueLok Elevate Transverse Bone Transport System is a modular external fixation device designed for transverse bone transport. It promotes local vascular and wound healing through controlled corticotomy and gradual distraction. The system is intended for adult patients with bony and/or soft tissuedefects.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 years or older at the time of surgery Willing and able to sign and date the study-specific informed consent form in accordance with national and institutional ethics requirements Willing and able to comply with requirements of the protocol, including follow-up requirements Indicated for surgical intervention using the TrueLok Elevate Transverse Bone Transport System for the treatment of soft tissue defects in the form of lower limb ulcers

Presence of a chronic ulcer, defined as:

* Present for at least 3 months, and
* Unresponsive to standard non-surgical or surgical wound management, including but not limited to debridement, negative pressure wound therapy (VAC), offloading, antibiotics, or vascular optimisation

Exclusion Criteria:

Mental or cognitive impairment or physiological or behavioural conditions that, in the opinion of the investigator, would preclude reliable adherence to postoperative care instructions, follow-up assessments, or study procedures

Known or presenting with the following signs of a systemic inflammatory response syndrome (SIRS) as exhibiting two or more of the following conditions:

o

* Heart rate >90 beats/min
* Respiratory rate >20 breaths/min
* PaCO2 <32-mm Hg
* White blood cell count >12.000 or <4.000/cu mm
* 10% immature (band) forms Known hypersensitivity or allergy to any material used in the TrueLok Elevate Transverse Bone Transport System (e.g., stainless steel, titanium) Current participation in another interventional clinical study that, in the opinion of the investigator, may interfere with the objectives or outcomes of this study Presence of active malignancy or systemic infection that, in the investigator's opinion, may interfere with wound healing or the study protocol Life expectancy of less than 12 months Simultaneous bilateral application of the TrueLok Elevate Transverse Bone Transport System Current incarceration at the time of enrolment Any condition or clinical circumstance that, in the opinion of the investigator, would make participation not in the best interest of the subject or would interfere with the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by chronic foot ulcers
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2028-11-24 (Estimated); Study Completion 2028-11-24 (Estimated)

PRIMARY OUTCOMES:
Complete ulcer healing | 12 months
  Proportion of subjects achieving complete ulcer healing within 12 months of device removal. Healing is defined as full epithelialisation with no open wound.

CONTACTS AND LOCATIONS:
Locations (1):
- Helios Klinikum Wuppertal GmbH, Wuppertal, Germany